CLINICAL TRIAL: NCT05491460
Title: Study on the Pharmacokinetics and Point of Care Testing After a Single Dose of 150 mg Dabigatran, 20 mg Rivaroxaban, 5 mg Apixaban, and 60 mg Edoxaban in Healthy Male Subjects
Brief Title: Pharmacokinetics and Point of Care Testing of Direct Oral Anticoagulants Subjects
Acronym: PHAPOCU
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Doasense GmbH (Industry)
Responsible Party: Principal Investigator, Job Harenberg, Clinical Professor, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PhaKiDo-001
Record Dates: First submitted 2019-02-11; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Anticoagulant Therapy
Keywords: anticoagulant; direct oral anticoagulant; apixaban; edoxaban; rivaroxaban; dabigatran; coagulation; point of care method
MeSH Terms: conditions — Thrombosis | interventions — apixaban; edoxaban; Dabigatran; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Apixaban (Active Comparator): Volunteers receive one oral dose of 5mg Apxiaban followed by sequential blood and urine sampling over 72 hours During the study liquid-chromatography mass-spectrometry analysis is performed in plasma and urine and DOAC Dipstick in urine.
  Biological and clinical safety parameters are measured.
  Interventions: Drug: Apixaban 5 MG Tab
- Dabigatran (Active Comparator): Volunteers receive one oral dose of 150mg Dabigatran followed by sequential blood and urine sampling over 72 hours During the study liquid-chromatography mass-spectrometry analysis is performed in plasma and urine and DOAC Dipstick in urine.
  Biological and clinical safety parameters are measured.
  Interventions: Drug: Dabigatran 150 MG Tab
- Edoxaban (Active Comparator): Volunteers receive one oral dose of 60mg Edoxaban followed by sequential blood and urine sampling over 72 hours During the study liquid-chromatography mass-spectrometry analysis is performed in plasma and urine and DOAC Dipstick in urine.
  Biological and clinical safety parameters are measured.
  Interventions: Drug: Edoxaban 60Mg Tab
- Rivaroxaban (Active Comparator): Volunteers receive one oral dose of 20mg Rivaroxaban followed by sequential blood and urine sampling over 72 hours During the study liquid-chromatography mass-spectrometry analysis is performed in plasma and urine and DOAC Dipstick in urine.
  Biological and clinical safety parameters are measured.
  Interventions: Drug: Rivaroxaban 20 MG Tab

INTERVENTIONS:
Drug: Apixaban 5 MG Tab — oral intake
  Other Names: Edoxaban, Dabigatran, rivaroxaban
  Arms: Apixaban
Drug: Dabigatran 150 MG Tab — oral intake
  Other Names: Apixaban, Edoxaban, Rivaroxaban
  Arms: Dabigatran
Drug: Edoxaban 60Mg Tab — oral intake
  Other Names: Apixaban, Dabigatran, Rivaroxaban
  Arms: Edoxaban
Drug: Rivaroxaban 20 MG Tab — oral intake
  Other Names: Apixaban, Edoxaban, Dabigatran
  Arms: Rivaroxaban

SUMMARY:
DOACs are increasingly used since 8 years. Standard coagulation tests (Prothrombin time [PT] and activated partial thromboplastin time [aPTT]) from plasma samples show a high variation. Special coagulation tests like hemoclot for dabigatran and chromogenic substrate assays for Rivaroxaban, Apixaban, and Edoxaban are time-consuming and can be performed only in specialized laboratories. In specific medical situations like in patients such as emergency procedures, stroke (before starting thrombolytic therapy), trauma, general surgery or other invasive procedures, it may be necessary for medical decision making to know the presence or absence of a DOAC in patient's body fluid. Until now there is no rapid, specific and sensitive coagulation test available in the market.

DETAILED DESCRIPTION:
This prospective, open-label, controlled, not randomized trial in healthy volunteers to investigate comparatively the pharmacokinetics of the direct oral anticoagulants in plasma and in urine with LC-MS/MS and in urine by DOAC Dipstick.

ELIGIBILITY:
Inclusion Criteria:

* Fully signed and dated written informed consent

  * Age >18 years
  * healthy

Exclusion Criteria:

* Patients not able to provide urine samples.

  * Patients not able to understand the informed consent or severe mentally disabled.
  * Patients in the end-stage of a severe disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 24 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy and specificity of the DOAC Dipstick compare to LC-MSMS | up to 6 months
  Assess the accuracy and specificity of the IVD for oral direct factor Xa and thrombin inhibitors from urine samples of patients True positive and true negative rate of the point of care test (POCT) by comparison with the results obtained by bioanalytical quantification

SECONDARY OUTCOMES:
Comparison of qualitative POCT with quantitative LC-MS/MS | up to 6 months
  Comparison of qualitative POCT with quantitative LC-MS/MS Investigator readings of POCT test results as compared to LC-MS/MS
Questionnaire on handling and usability | up to 6 months
  Specific questions to be answered using Lickert scale by personal performing the test

CONTACTS AND LOCATIONS:
Overall Officials: Armin Schultz, MD, Study Director — Clinical Research Services
Locations (1):
- Clincial Research Serivces, Mannheim, Germany

REFERENCES:
- [Background] Harenberg J, Schreiner R, Hetjens S, Weiss C. Detecting Anti-IIa and Anti-Xa Direct Oral Anticoagulant (DOAC) Agents in Urine using a DOAC Dipstick. Semin Thromb Hemost. 2019 Apr;45(3):275-284. doi: 10.1055/s-0038-1668098. Epub 2018 Aug 22. PMID 30134449